CLINICAL TRIAL: NCT00214383
Title: Internet Telehealth for Pediatric Asthma Case Management
Acronym: CHESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002-163; 5R01NR007889-02 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Asthma
Keywords: pediatric asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHESS + Case Mgt (Experimental): Case Management (with monthly support calls) and CHESS services were available for a 12 month intervention period. Support calls refer to check in calls by a nurse to the parents to see how the child is doing. CHESS services include access to a website with information on asthma management, discussion groups and a case manager. The website also include a management tool for asthma symptoms check in, and the case manager used the information entered to tailor the homepage to individual clients.
  Interventions: Behavioral: CHESS Internet telehealth
- Control (No Intervention): Control-usual care. Usual care refers to the manner in which clients generally manage their asthma.

INTERVENTIONS:
Behavioral: CHESS Internet telehealth — CHESS Internet telehealth
  Arms: CHESS + Case Mgt

SUMMARY:
The original and primary aim of this study is to evaluate the effects of CHESS with Nurse Case Management on asthma control (symptom-free days), and adherence factors of children aged 4-12. The investigators have expanded the scope of the specific aims. The criteria for their expanded aim is to also interview low-income African-American caregivers to gain an understanding of how they conceptualize their child's asthma, and what they consider to be barriers or facilitators to managing their child's asthma. There is no change in the investigators' original aim.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children, aged 4-12 with moderate to severe asthma

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 301 (Actual)
Dates: Start 2004-05; Primary Completion 2007-08 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Gustafson, PhD, Principal Investigator — University of Wisconsin, Madison

REFERENCES:
- [Background] Wise M, Gustafson DH, Sorkness CA, Molfenter T, Staresinic A, Meis T, Hawkins RP, Shanovich KK, Walker NP. Internet telehealth for pediatric asthma case management: integrating computerized and case manager features for tailoring a Web-based asthma education program. Health Promot Pract. 2007 Jul;8(3):282-91. doi: 10.1177/1524839906289983. Epub 2006 Aug 23. PMID 16928987
- [Result] Wise M, Pulvermacher A, Shanovich KK, Gustafson DH, Sorkness C, Bhattacharya A. Using action research to implement an integrated pediatric asthma case management and eHealth intervention for low-income families. Health Promot Pract. 2010 Nov;11(6):798-806. doi: 10.1177/1524839909334621. Epub 2009 Jun 10. PMID 19515862
- [Result] Gustafson D, Wise M, Bhattacharya A, Pulvermacher A, Shanovich K, Phillips B, Lehman E, Chinchilli V, Hawkins R, Kim JS. The effects of combining Web-based eHealth with telephone nurse case management for pediatric asthma control: a randomized controlled trial. J Med Internet Res. 2012 Jul 26;14(4):e101. doi: 10.2196/jmir.1964. PMID 22835804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study extended 1,988 invitations, resulting in eligibility screening for 702 cases over the phone. A total of 305, or about 15% of the 1,988 invitations, enrolled. Some of the reasons for non-enrollment include inability of clients to reach phone, not having moderate to severe asthma, or up to 3 no shows for scheduled intake appointments.
Pre-assignment Details: After initial eligibility screening, 305 parent/child dyads enrolled for study. However, four dyads dropped out after intake, but prior to randomization. Of the remaining dyads, 153 were assigned to the control group and 148 to the experimental group.
Groups:
- CHESS + Case Mgt: Case Management (with monthly support calls) and CHESS services were available for a 12 month intervention period.
- Control: Control-usual care
Period: Overall Study
Arm/Group | CHESS + Case Mgt | Control
Started | 148 | 153
Completed | 132 | 127
Not Completed | 16 | 26
Not completed — Lost to Follow-up | 16 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHESS + Case Mgt | Control | Total
Number analyzed (Participants) | 148 | 153 | 301
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 148 | 153 | 301
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.65 (2.61) | 8.18 (2.45) | 7.92 (2.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 66 | 117
  Male | 97 | 87 | 184
Region of Enrollment [Number; unit: participants]
  United States | 148 | 153 | 301

OUTCOME MEASURES:

1. Primary Outcome: Percentage Changed in Adherence Score
Description: A baseline number of participants less dropouts was gauged against the weighted average of the number of participants in study period. The percentage change in adherence from baseline through the study was measured and is reported below, together with confidence intervals.
Time Frame: Baseline compared to the mean of the combined 3, 6, 9, and 12 month scores
Population: Forty two dyads dropped out after randomization. Of these, 16 were from the experimental group and 26 from the control group.
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | CHESS + Case Mgt | Control
Number analyzed (Participants) | 132 | 127
Percent change | 2.06 [-4.74 to 8.86] | .58 [-6.24 to 7.40]

2. Primary Outcome: Number of Symptom-free Days
Description: A comparison in the average number of days that a child goes without asthma symptoms between experimental and control groups are shown below.
Time Frame: Baseline compared to the mean of the combined 3, 6, 9, and 12 month scores
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | CHESS + Case Mgt | Control
Number analyzed (Participants) | 132 | 127
Days | 1.38 [1.12 to 1.71] | 1.26 [.98 to 1.61]

3. Secondary Outcome: Improvement in Asthma Control
Description: A six item survey on a seven point Likert scale measuring daytime and nocturnal asthma symptoms, missed school days and rescue medication use in the previous seven days. Lower scores signal better asthma control.
Time Frame: Baseline compared to the mean of the combined 3, 6, 9, and 12 month scores
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Likert scale
Arm/Group | CHESS + Case Mgt | Control
Number analyzed (Participants) | 132 | 127
Likert scale | -.42 [-.60 to -.25] | -.11 [-.29 to .07]

ADVERSE EVENTS:
Arm/Group | CHESS + Case Mgt | Control
Serious Adverse Events (participants affected / at risk) | 0/148 | 0/153
Other Adverse Events (participants affected / at risk) | 0/148 | 0/153

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No